CLINICAL TRIAL: NCT02939144
Title: An Investigation Into the Effect of Liquorice Ingestion on the Salivary Cortisol to Cortisone Molar Ratio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016LAB86
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Apparent Mineralocorticoid Excess
MeSH Terms: conditions — Mineralocorticoid Excess Syndrome, Apparent | interventions — Glycyrrhiza glabra extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liquorice (Experimental): Participants of the single-arm study will ingest liquorice candy and their blood, saliva and urine samples will be collected. They will be regularly monitored for any potential side effects.
  Interventions: Dietary Supplement: Liquorice

INTERVENTIONS:
Dietary Supplement: Liquorice — Liquorice ingestion will mimic the inherited condition of 'Apparent mineralocorticoid excess (AME)by showing the effects of the reduced activity of 11ßHSD-2 (which leads to an accumulation of cortisol which binds MR and hence has the effect of aldosterone).

SUMMARY:
Aldosterone, the major mineralocorticoid hormone and cortisol, the major glucocorticoid hormone are produced in the adrenal gland. Aldosterone binds intracellular mineralocorticoid receptors (MR) in the kidney promoting urinary reabsorption of sodium and water and excretion of potassium and hydrogen ions. Unregulated mineralocorticoid excess may, therefore, lead to high blood pressure due to sodium and water retention and hypokalaemic alkalosis.

Blood concentrations of cortisol which has equal affinity for MR are 1000fold greater than those of aldosterone. Therefore in order not to overwhelm MR, cortisol needs to be inactivated before it binds MR. This is achieved by the enzyme 11-betahydroxysteroid dehydrogenase type 2 (11ßHSD-2) in the kidney which rapidly inactivates cortisol to cortisone (this process allows only aldosterone to bind MR). Reduced activity of 11ßHSD-2 leads to an accumulation of cortisol which binds MR and hence has the effect of aldosterone. Reduced activity of 11ßHSD-2 may be seen in the inherited condition of 'Apparent mineralocorticoid excess (AME)' or in excessive liquorice ingestion. The diagnosis of AME and liquorice toxicity is difficult due to unavailability of diagnostic urine analysis in most general laboratories. Cortisol in the salivary glands, similarly to that in kidneys, is metabolised by 11β-HSD2 to cortisone. It is proposed that increased salivary cortisol/cortisone ratio could offer a simple and convenient diagnostic test for AME and liquorice toxicity and can be used as a surrogate marker of urinary cortisol/cortisone ratio. The advantages of salivary cortisol/cortisone include non-invasiveness making it stress free for the patient, no risk of needle stick injury and ease of collection allowing potential home testing and posting of samples.

DETAILED DESCRIPTION:
Twelve healthy normotensive individuals, between 20-65 years old, without high blood pressure will be recruited to the study. Study individuals will be recruited among the hospital staff on a voluntary basis.

The study period will consist of three phases prior to which potential volunteers will be identified:

* Phase 1: Run-in week with definition of baseline values.
* Phase 2: Six day period with a daily intake of 550 mg of Glycyrrhizin for 5 days in the form of liquorice confectionary.
* Phase 3: Two week washout period.

Phase 1: The run-in week:

* Potential volunteers will be identified and given study information (participant information sheet) allowing time to consider taking part. Most volunteers to be recruited among the hospital staff.
* Written consent will be obtained from volunteers by study investigators.
* Volunteers will have their blood pressure, weight and height checked and will be assessed for inclusion and exclusion criteria.
* The office blood pressure will be measured after 5 min rest. Blood pressure will be measured on two different days during the run-in period, twice each time, and the mean of these four measurements will be used as the baseline value.
* Baseline samples (taken any day within the run-in week; days -6, -5, -4, -3,-2,-1, 0):

  * Saliva samples on two consecutive days between 08.30h to 09.30h.
  * One blood sample between 08.30h to 09.30h.
  * One 24h urine sample.

Phase 2: A six day study period (days 1, 2, 3, 4, 5, 6):

* Twelve volunteers will ingest confectionary liquorice containing 550 mg of Glycyrrhizin in divided amounts each day for five days. The liquorice, in the form of sugar-free candies, will be ingested three times per day at least 30 minutes prior to meals in the morning, afternoon and evening.
* Volunteers will be requested to refrain from eating grapefruit or drinking grapefruit juice during the study period.
* The liquorice candies will be weighed to give the correct dose of glycyrrhizin.
* Subjects will be clinically monitored daily during liquorice consumption for any potential side effects, including headaches, swelling, dyspepsia, dizziness, joint pain, muscle aches, and palpitations.
* Office blood pressure, heart rate and weight will be measured daily during liquorice consumption.
* Volunteers will collect salivary samples daily between 08.30h to 09.30h for six days.
* A blood sample will be collected on day 6 between 8.30h to 09.30h.
* A 24h urine sample will then be collected on starting at 8.30h to 09.30h and completed on 8.30h to 09.30h on day 7.

Phase 3: At the end of a two week washout period (Day 19):

* Salivary and blood samples will be collected between 08.30h to 09.30h
* A 24h urine sample will then be collected starting at 8.30h to 09.30h on day 19 and completed on 8.30h to 09.30h on day 20.
* Office blood pressure, pulse rate and weight will recorded.

In total 40 mls of saliva, 30 mls blood and three 24h urine samples will be collected. Labelling of saliva, blood and urine samples will be anonymized. Saliva and blood samples will be centrifuged. The separated serum/plasma and extracted saliva will be kept frozen at -80oC until analysed in one batch (to minimise analytical variation). 24h urine samples will have their volume measured and an aliquot will be kept frozen at -80oC until analysed in one batch.

ELIGIBILITY:
Inclusion Criteria:

* Normal blood pressure without electrolyte abnormalities.
* Healthy, without any known medical conditions or treatment other than the contraceptive pill.

Exclusion Criteria:

* Pregnant women.
* Subjects with learning disability or those lacking mental capacity to give consent.
* On prescribed and over-the-counter medication and herbal remedies excluding the contraceptive pill.
* Any known medical condition.
* Subjects with difficult blood access.
* Subjects with dental disease.
* Those using tobacco in any form.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

PRIMARY OUTCOMES:
salivary cortisol/cortisone ratio induced by liquorice (glycyrrhetinic acid and its metabolites) ingestion | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rousseau Gama, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No